CLINICAL TRIAL: NCT00874848
Title: Efficacy and Safety Study of Imprime PGG® Injection in Combination With Cetuximab and Concomitant Paclitaxel and Carboplatin Therapy in Patients With Previously Untreated Advanced (Stage IIIB or IV) Non-Small Cell Lung Cancer
Brief Title: Efficacy/Safety of Imprime PGG With Cetuximab & Paclitaxel/Carboplatin Therapy in Pts With Untreated Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HiberCell, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BT-CL-PGG-LCA0822
Record Dates: First submitted 2009-04-01; First posted 2009-04-03 (Estimated); Results first posted 2016-11-29 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-10

CONDITIONS: NSCLC
Keywords: Imprime PGG; NSCLC; Cetuximab
MeSH Terms: interventions — Cetuximab; Paclitaxel; Albumin-Bound Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Imprime PGG (Experimental): Imprime PGG Injection + Cetuximab + Paclitaxel/Carboplatin
  Interventions: Biological: Imprime PGG Injection; Biological: Cetuximab; Drug: Paclitaxel; Drug: Carboplatin
- Control (Active Comparator): Cetuximab + Paclitaxel/Carboplatin
  Interventions: Biological: Cetuximab; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Biological: Imprime PGG Injection — 4 mg/kg i.v. over 2 hrs, weekly, in three week cycles
  Arms: Imprime PGG
Biological: Cetuximab — initial loading dose of 400 mg/m^2 over 120 min and subsequent doses at 250 mg/m^2 over 60 min, weekly on Days 1, 8 and 15 of each 3-week treatment cycle
  Other Names: Erbitux
Drug: Paclitaxel — 200 mg/m^2 i.v. over 3 hr on Day 2 of each 3-week treatment cycle for the first 4 to 6 treatment cycles
  Other Names: Abraxane; Taxol; Onxol; Nov-Onxol
Drug: Carboplatin — dose equal to an AUC of 6 mg/mL · min based on the Calvert formula; i.v. over 30 min on Day 2 of each 3-week treatment cycle for the first 4 to 6 treatment cycles
  Other Names: Paraplatin

SUMMARY:
The Phase 2 study described in this protocol will serve to evaluate the antitumor activity, safety and pharmacokinetic profile of Imprime PGG when combined with cetuximab and concomitant paclitaxel and carboplatin therapy in patients with previously untreated advanced NSCLC. Additionally, this study will provide guidance for the design of more definitive efficacy studies of Imprime PGG in NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Has read, understood and signed the informed consent form (ICF) approved by the Independent Review Board/Ethics Committee (IRB/EC)
2. Is between the ages of 18 and 75 years old, inclusive
3. Has histologically or cytologically confirmed stage IIIB (malignant pericardial or pleural effusion) or stage IV non-small cell lung cancer
4. Has measurable disease, defined as at least one tumor that fulfills the criteria for a target lesion according to RECIST
5. Has an ECOG performance status of 0 or 1
6. Has a life expectancy of > 3 months
7. Has adequate hematologic function as evidenced by:

   * ANC ≥ 1,500/μL
   * PLT ≥ 100,000/μL
   * HGB ≥ 9 g/dL obtained within 1 week prior to the first dose of study medication;
8. Has adequate renal function as evidenced by:

   * Serum creatinine ≤ 1.5 X the upper limit of normal (ULN) for the reference lab
   * Urine dipstick for proteinuria of < 1+ (i.e., either 0 or trace) within 2 weeks of Day 1 If urine dipstick is ≥ 1+, then urine protein excretion must be ≤ 500 mg over a 24 hour collection obtained within 1 week prior to the first dose of study medication;
9. Has adequate hepatic function as evidenced by:

   * Serum total bilirubin ≤ 1.0 mg/dL
   * AST ≤ 2.5X ULN for the reference lab (≤ 5X ULN for subjects with known hepatic metastases)
   * ALT ≤ 2.5X ULN for the reference lab (≤ 5X ULN for subjects with known hepatic metastases) obtained within 1 week prior to the first dose of study medication;
10. If a woman of childbearing potential or a fertile man (and his partners), must agree to use an effective form of contraception (hormonal contraceptive, double-barrier method or abstinence) during the study.

Exclusion Criteria:

1. Has received prior systemic chemotherapy at any time for lung cancer;
2. Has received previous radiation therapy to >30% of active bone marrow or any radiation therapy within 3 weeks of Day 1
3. Has a known hypersensitivity to baker's yeast, or has an active yeast infection
4. Has had previous exposure to Betafectin® or Imprime PGG
5. Has an active infection
6. Presents with any of the following medical diagnoses/conditions at the time of screening:

   * Central nervous system (CNS) metastases
   * Uncontrolled hypertension (>150/100 mmHg) or hypertension that requires > two agents for adequate control
   * Peripheral neuropathy ≥ grade 2 from any cause
   * Fever of >38.5° C within 3 days prior to screening or Day 1, initial dosing
   * Known HIV/AIDs, Hepatitis B, Hepatitis C, connective tissue or autoimmune disease, or other clinical diagnosis, ongoing or intercurrent illness that in the physician's opinion could interfere with participation
7. Has a history of any of the following medical diagnoses/conditions:

   * Myocardial infarction or an unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure) within the previous 6 months
   * Second malignancy within the previous 5 years, other than basal cell carcinoma, cervical intra-epithelial neoplasia or curatively treated prostate cancer with a PSA of <2.0 ng/mL
8. Has a known hypersensitivity to cetuximab, murine proteins, or any component of cetuximab
9. Has a know sensitivity to Cremophor EL
10. Has previously received treatment with cetuximab
11. If female, is pregnant or breast-feeding
12. Is receiving concurrent investigational therapy or has received investigational therapy within a period of 30 days prior to the first scheduled day of dosing (investigational therapy is defined as treatment for which there is currently no regulatory-authority-approved indication)
13. Has previously received an organ or progenitor/stem cell transplant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-08; Primary Completion 2012-11 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Folker Schneller, MD, Principal Investigator — Technical University, Munich
Locations (14):
- United States (5):
  - Medical College of Georgia, Augusta, Georgia
  - Providence Medical Group, Terre Haute, Indiana
  - University of Minnesota, Minneapolis, Minnesota
  - Mary Crowley Medical Research Center, Dallas, Texas
  - Allison Cancer Center, Midland, Texas
- Germany (9):
  - Helios Clinic Emil von Behring, Berlin
  - Municipal Clinic Frankfurt Hoescht, Frankfurt
  - Georg-August University Gottingen, Göttingen
  - University Clinical Heidelberg, Heidelberg
  - Clinic Minden, Minden
  - Techincal University of Munich, Munich
  - Clinic Nurnberg Nord, Nuremberg
  - Universitätsklinikum Ulm, Ulm
  - HELIOS Klinikum Wuppertal, Medizinische Klinik 1, Wuppertal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thomas M, Sadjadian P, Kollmeier J, Lowe J, Mattson P, Trout JR, Gargano M, Patchen ML, Walsh R, Beliveau M, Marier JF, Bose N, Gorden K, Schneller F 3rd. A randomized, open-label, multicenter, phase II study evaluating the efficacy and safety of BTH1677 (1,3-1,6 beta glucan; Imprime PGG) in combination with cetuximab and chemotherapy in patients with advanced non-small cell lung cancer. Invest New Drugs. 2017 Jun;35(3):345-358. doi: 10.1007/s10637-017-0450-3. Epub 2017 Mar 16. PMID 28303530

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A randomized, Simon 2-stage flexible design with 22 patients enrolled in stage 1 and 68 additional patients in stage 2, for a total of 90 subjects (60 in the Imprime PGG arm and 30 in the Control arm) enrolled competitively across US and German clinical sites.
  First subject enrolled: 17 Aug 2009 Last subject last visit: 15 Nov 2012
Pre-assignment Details: A total of 90 participants enrolled, 88 participants received at least one dose of study treatment, and 2 participants did not receive any study treatment.
Groups:
- Imprime PGG Arm: Imprime PGG® infusion:
  4 mg/kg i.v. over 2 to 4 hrs on Days 1, 8 and 15 of each 3-week treatment cycle;
  Cetuximab infusion:
  initial loading dose of 400 mg/m2 over 120 min and subsequent doses at 250 mg/m2 over 60 min, on Days 1, 8 and 15 of each 3-week treatment cycle;
  Paclitaxel infusion:
  200 mg/m2 i.v. over 3 hr on Day 2 of each 3-week treatment cycle for the first 4 to 6 treatment cycles
  Carboplatin infusion:
  dose equal to an AUC of 6 mg/mL · min based on the Calvert formula; i.v. over 30 min on Day 2 of each 3-week treatment cycle for the first 4 to 6 treatment cycles.
  Following the completion of at least the initial 4 treatment cycles (but no more than 6), participants experiencing stable disease, or a complete or partial response, were eligible to discontinue the chemotherapy treatment and continue dosing of Imprime PGG and cetuximab for a maximum of 18 treatment cycles without a treatment extension being authorized by the Sponsor.
- Control Arm: Cetuximab infusion:
  initial loading dose of 400 mg/m2 over 120 min and subsequent doses at 250 mg/m2 over 60 min, on Days 1, 8 and 15 of each 3-week treatment cycle;
  Paclitaxel infusion:
  200 mg/m2 i.v. over 3 hr on Day 2 of each 3-week treatment cycle for the first 4 to 6 treatment cycles
  Carboplatin infusion:
  dose equal to an AUC of 6 mg/mL · min based on the Calvert formula; i.v. over 30 min on Day 2 of each 3-week treatment cycle for the first 4 to 6 treatment cycles.
  Following the completion of at least the initial 4 treatment cycles (but no more than 6), participants experiencing stable disease, or a complete or partial response, were eligible to discontinue the chemotherapy treatment and continue dosing of cetuximab for a maximum of 18 treatment cycles without a treatment extension being authorized by the Sponsor.
Period: Overall Study
Arm/Group | Imprime PGG Arm | Control Arm
Started | 59 | 29
Discontinued | 59 | 28
Completed | 0 (Pts who completed 18 tx cycles without progressive disease were defined as completing treatment.) | 1 (Pts who completed 18 tx cycles without progressive disease were defined as completing treatment.)
Not Completed | 59 | 28
Not completed — Adverse Event | 13 | 2
Not completed — Progressive neoplastic disease | 38 | 18
Not completed — Withdrawal by Subject | 7 | 4
Not completed — Noncompliance | 1 | 1
Not completed — Failure to comply with protocol | 0 | 1
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Population: The safety population comprised all randomized participants who received any amount of Imprime PGG, cetuximab, paclitaxel or carboplatin.
Groups:
- Imprime PGG Arm: Imprime PGG Injection + Cetuximab + Paclitaxel/Carboplatin
- Control Arm: Cetuximab + Paclitaxel/Carboplatin
- Total: Total of all reporting groups
Arm/Group | Imprime PGG Arm | Control Arm | Total
Number analyzed (Participants) | 59 | 29 | 88
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.3 (9.45) | 62.4 (7.04) | 60.45 (8.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 27
  Male | 44 | 17 | 61
Race/Ethnicity, Customized [Number; unit: participants]
  White | 56 | 29 | 85
  Black | 2 | 0 | 2
  Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 2 | 6
  Germany | 55 | 27 | 82
ECOG [Number; unit: participants] — ECOG Score: runs from 0 to 5, with 0 denoting perfect health and 5 death.
  0 - Asymptomatic (Fully active, able to carry on all predisease activities without restriction)
  1 - Symptomatic but completely ambulatory (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature. For example, light housework, office work)
  participants
    Score = 0 | 20 | 10 | 30
    Score = 1 | 38 | 18 | 56
    Missing | 1 | 1 | 2
Baseline Height [Mean (Standard Deviation); unit: cm] | 171.1 (7.51) | 170.0 (8.90) | 170.8 (7.96)
Baseline Weight [Mean (Standard Deviation); unit: kg] | 76.2 (16.52) | 72.8 (12.19) | 75.0 (15.24)
Baseline Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.9 (4.95) | 25.1 (3.00) | 25.6 (4.40)
Time from Initial Tumor Diagnosis [Mean (Standard Deviation); unit: months] | 0.9 (1.04) | 0.9 (1.53) | 0.9 (1.21)
Prior Cancer Treatment [Number; unit: participants]
  Radiotherapy | 0 | 3 | 3
  Surgery | 23 | 13 | 36
  Chemotherapy | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) in Each Study Arm Based on Independent Central Radiology Review
Description: Overall objective response rate was defined as the number of participants experiencing a best overall response of either complete response (CR) or partial response (PR) based on the modified RECIST v1.0 criteria.
  The analysis performed for this study utilized a modified RECIST v1.0 in which a confirmed response after the initial response assessment was not required by repeat assessment. With the use of centrally read, blinded radiological assessments performed by independent radiologists, and the use of randomization between study arms, the criterion requiring a 'confirmation' response was removed. All other RECIST v1.0 criteria remained unmodified and implemented as stated in the guidelines.
Time Frame: From first dose to disease progression or last tumor assessment before treatment discontinuation due to any reason, up to 15 months
Population: The primary efficacy population comprised all randomized subjects who had no major violations of inclusion/exclusion or significant protocol violations & received any amount of cetuximab, paclitaxel or carboplatin therapy or Imprime PGG, & had an evaluable baseline scan & at least one evaluable post-baseline response based on modified RECIST v1.0.
Measure: Number; unit: participants
Arm/Group | Imprime PGG Arm | Control Arm
Number analyzed (Participants) | 41 | 26
participants
  Number of participants with best response of CR | 0 | 0
  Number of participants with best response of PR | 15 | 6
Statistical Analysis 1: Comparison: Imprime PGG Arm vs Control Arm; Test type: Superiority or Other; p = 0.2895, Fisher Exact

2. Secondary Outcome: Overall Survival (OS) in Each Study Arm Based on the Safety Population
Description: Overall survival (OS) was defined as the time from the date of randomization until the date of documented death of the subject due to any cause, including death due to relapses that were successfully retreated. Subjects who were lost to follow-up or who were still alive at the time of analysis were censored at the last contact dates.
Time Frame: From the time of randomization to death, subject being lost to follow-up or study completion
Population: The safety population comprised all randomized subjects who received any amount of Imprime PGG, cetuximab, paclitaxel or carboplatin.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Imprime PGG Arm | Control Arm
Number analyzed (Participants) | 59 | 29
months | 10.3 [8.6 to 15.1] | 12.4 [9.3 to 17.4]

3. Secondary Outcome: Disease Control Rate (DCR) in Each Study Arm Based on Independent Central Radiology Review
Description: The disease control rate (DCR) was defined as the number of participants experiencing a best overall tumor response of either CR, PR or SD. For stable disease (SD), follow-up measurements must have met the SD criteria at least once after study entry at a minimum interval of 6 weeks.
  The analysis performed for this study utilized a modified RECIST v1.0 in which a confirmed response after the initial response assessment was not required by repeat assessment. With the use of centrally read, blinded radiological assessments performed by independent radiologists, and the use of randomization between study arms, the criterion requiring a 'confirmation' response was removed. All other RECIST v1.0 criteria remained unmodified and implemented as stated in the guidelines.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Imprime PGG Arm | Control Arm
Number analyzed (Participants) | 41 | 26
participants | 35 | 21

4. Secondary Outcome: Complete Response (CR), Partial Response (PR), and Stable Disease (SD) Rates in Each Study Arm Based on Independent Central Radiology Review
Description: The best observed overall response rates were defined as the number of participants experiencing a best overall response of either complete response (CR), partial response (PR) or stable disease (SD) based on the modified RECIST v1.0 criteria. For stable disease (SD), follow-up measurements must have met the SD criteria at least once after study entry at a minimum interval of 6 weeks.
  The analysis performed for this study utilized a modified RECIST v1.0 in which a confirmed response after the initial response assessment was not required by repeat assessment. With the use of centrally read, blinded radiological assessments performed by independent radiologists, and the use of randomization between study arms, the criterion requiring a 'confirmation' response was removed. All other RECIST v1.0 criteria remained unmodified and implemented as stated in the guidelines.
Time Frame: From the first dose to disease progression or last tumor assessment before treatment discontinuation due to any reason, up to 15 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Imprime PGG Arm | Control Arm
Number analyzed (Participants) | 41 | 26
participants
  Number of participants with best response of CR | 0 | 0
  Number of participants with best response of PR | 15 | 6
  Number of participants with best response of SD | 20 | 15

5. Secondary Outcome: Duration of Objective Tumor Response in Each Study Arm Based on Independent Central Radiology Review
Description: The duration of objective tumor response was measured from the time at which criteria are met for CR or PR (whichever status is recorded first) until the first date on which recurrence or progressive disease is objectively documented per modified RECIST v1.0. Subjects who did not progress as of the data cutoff date were censored at their last tumor assessment date.
  The analysis performed for this study utilized a modified RECIST v1.0 in which a confirmed response after the initial response assessment was not required by repeat assessment. With the use of centrally read, blinded radiological assessments performed by independent radiologists, and the use of randomization between study arms, the criterion requiring a 'confirmation' response was removed. All other RECIST v1.0 criteria remained unmodified and implemented as stated in the guidelines.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Imprime PGG Arm | Control Arm
Number analyzed (Participants) | 15 | 6
months | 4.4 [2.8 to 6.5] | 4.1 [1.4 to 5.4]

6. Secondary Outcome: Duration of Time to Progression (TTP) in Each Study Arm Based on Independent Central Radiology Review
Description: Time-to-progression (TTP) was defined as the time from the date of randomization to the first date of documented progressive disease. Progressive disease was identified by radiologic progressive disease according to modified RECIST v1.0, or in the case of the Investigator Radiologic Review, it may also be defined by clinical progression as determined by the investigator.
  If a subject received any further anti-cancer therapy without prior documentation of disease progression, the subject was censored at the date of last tumor assessment before starting anti-cancer treatment. Subjects who died on study from other causes (not related to study disease) and subjects who were lost to follow-up or who were alive without documented progressive disease as of the data cut-off date for analysis were censored at the last tumor assessment date.
Time Frame: From time of randomization to first date of documented progression, or last tumor assessment date, up to 15 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Imprime PGG Arm | Control Arm
Number analyzed (Participants) | 41 | 26
months | 6.4 [4.3 to 8.3] | 6.0 [4.3 to 7.1]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the first dose of investigational product to the discontinuation of study plus 30 days after the last dose of study drug or until the subject began alternative therapy.
Arm/Group | Imprime PGG Arm | Control Arm
Serious Adverse Events (participants affected / at risk) | 37/59 | 12/29
Other Adverse Events (participants affected / at risk) | 59/59 | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Imprime PGG Arm (N=59) | Control Arm (N=29)
Neutropenia (Blood and lymphatic system disorders) | 1 | 2
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Hypertrophic cardiomyopathy (Cardiac disorders) | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Death (General disorders) | 1 | 0
Disease progression (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 0
Infusion site extravasation (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Anaphylactic shock (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 1
Anal abscess (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Vascular occulsion (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Imprime PGG Arm (N=59) | Control Arm (N=29)
Neutropenia (Blood and lymphatic system disorders) | 22 | 14
Leukopenia (Blood and lymphatic system disorders) | 13 | 9
Anaemia (Blood and lymphatic system disorders) | 4 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 4
Tachycardia (Cardiac disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 25 | 12
Diarrhoea (Gastrointestinal disorders) | 24 | 9
Constipation (Gastrointestinal disorders) | 11 | 10
Vomiting (Gastrointestinal disorders) | 11 | 5
Abdominal pain (Gastrointestinal disorders) | 5 | 4
Stomatitis (Gastrointestinal disorders) | 4 | 4
Dyspepsia (Gastrointestinal disorders) | 4 | 2
Dysphagia (Gastrointestinal disorders) | 4 | 2
Abdominal pain upper (Gastrointestinal disorders) | 4 | 1
Flatulence (Gastrointestinal disorders) | 3 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 2
Fatigue (General disorders) | 30 | 17
Mucosal inflammation (General disorders) | 13 | 6
Chest pain (General disorders) | 10 | 5
Chills (General disorders) | 8 | 4
Pyrexia (General disorders) | 4 | 8
Oedema peripheral (General disorders) | 5 | 5
Asthenia (General disorders) | 3 | 3
General physical health deterioration (General disorders) | 3 | 2
Chest discomfort (General disorders) | 1 | 3
Hypersensitivity (Immune system disorders) | 3 | 3
Nasopharyngitis (Infections and infestations) | 6 | 3
Paronychia (Infections and infestations) | 6 | 2
Bronchitis (Infections and infestations) | 3 | 2
Cystitis (Infections and infestations) | 3 | 2
Folliculitis (Infections and infestations) | 5 | 0
Infection (Infections and infestations) | 3 | 0
Pneumonia (Infections and infestations) | 3 | 0
Oral fungal infection (Infections and infestations) | 0 | 2
Rhinitis (Infections and infestations) | 0 | 2
Haemoglobin decreased (Investigations) | 5 | 0
Amylase increased (Investigations) | 3 | 1
Blood magnesium decreased (Investigations) | 4 | 0
Blood phosphorus decreased (Investigations) | 2 | 2
Weight decreased (Investigations) | 3 | 1
White blood cell count decreased (Investigations) | 0 | 3
Body temperature increased (Investigations) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 13 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Polyneuropathy (Nervous system disorders) | 16 | 9
Paraesthesia (Nervous system disorders) | 7 | 9
Dizziness (Nervous system disorders) | 8 | 6
Headache (Nervous system disorders) | 7 | 4
Dysgeusia (Nervous system disorders) | 5 | 5
Neuropathy peripheral (Nervous system disorders) | 5 | 1
Ageusia (Nervous system disorders) | 4 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 3
Insomnia (Psychiatric disorders) | 7 | 5
Sleep disorder (Psychiatric disorders) | 3 | 1
Renal pain (Renal and urinary disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 10
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 28 | 19
Alopecia (Skin and subcutaneous tissue disorders) | 22 | 13
Dermatitis (Skin and subcutaneous tissue disorders) | 12 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 4
Skin fissures (Skin and subcutaneous tissue disorders) | 11 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 2
Hypotension (Vascular disorders) | 4 | 1
Thrombosis (Vascular disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No